CLINICAL TRIAL: NCT04685824
Title: Visual Rehabilitation in Macular Degeneration: a Pilot Study on Biofeedback Training and Home-based Mobile Virtual-reality Stimulation
Brief Title: Visual Telerehabilitation in AMD Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rate not reached.
Sponsor: Michael Reber (Other)
Responsible Party: Sponsor-Investigator, Michael Reber, Principal Investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020410013068
Record Dates: First submitted 2020-12-15; First posted 2020-12-28 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Macular Degeneration
Keywords: Visual rehabilitation; Oculus Go; Virtual-reality; Biofeedback
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback Training (Active Comparator): * Biofeedback training (BFT): 1 sessions of 4 x 20 minutes blocks. Rest time of 5 minutes between blocks. 1 session per week for 4 weeks (4 sessions total).
  * 30 min daily reading at home for 4 weeks.
  Interventions: Device: Biofeedback Training
- Biofeedback Training + Immersive VR (Experimental): * Biofeedback training (BFT) [1 sessions of 4 x 20 minutes blocks. Rest time of 5 minutes between blocks], 1 session per week for 4 weeks (4 sessions total).
  * 30 min daily reading at home for 4 weeks
  * Immersive virtual-reality stimulation (IVR) [1 session of 3 blocks of 15 trials of 20 seconds each. Rest time is 1-2 minute(s) between blocks], 1 session every 2 days for 4 weeks (14 sessions total).
  Interventions: Device: Biofeedback Training; Device: Immersive Virtual-Reality

INTERVENTIONS:
Device: Biofeedback Training — Audiovisual stimulation
Device: Immersive Virtual-Reality — Audiovisual stimulation
  Arms: Biofeedback Training + Immersive VR

SUMMARY:
Following the degeneration of the macula and the loss of central vision, the patients naturally relocate the fixation point for high visual acuity peripherally, in an eccentric and healthy part of the retina (PRL), to compensate for visual impairments. However, in many cases, the PRL lands on a sub-optimal retinal area and becomes useless. Modern low-vision rehabilitation procedures for AMD patients include biofeedback training (BFT) to relocate the PRL to a healthy retinal patch and acquire better fixation skills. This study seeks to combine BFT with home-based immersive virtual-reality audiovisual stimulation and measure feasibility and potential effectiveness on oculomotor control and visual perception.

ELIGIBILITY:
Inclusion Criteria:

* Dry-AMD.
* BCVA > 20/160.
* Ability to follow the visual and auditory stimuli and training instructions.
* Auditory test positive at 50Hz 25-60dBHL.
* Home Wi-Fi access.

Exclusion Criteria:

* Wet AMD.
* Both eyes with media opacity that impairs microperimetry testing.
* Inability to perform during testing and training.
* Psychoactive drugs consumption.
* 3 consecutive VRISE scores < 25 at inclusion.
* History of vertigo or dizziness
* Prior vision rehabilitation interventions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of home-based IVR audiovisual stimulation | 18 months
  Feasibility objectives for our pilot study to be considered successful:
  1. Number of patients completing the stimulation protocol: ≥ 13 out of 16 patients (81%) per group.
  2. Number of IVR sessions performed by the patients to consider the stimulation protocol complete: ≥ 13 sessions out of 16 (81%).
  3. Number of consecutive virtual-reality induced symptoms and effects (VRISE) scores < 25: ≤ 3 per patient during the treatment period.
  4. Number of patient drop-outs due to cybersickness (discomfort symptoms experienced in VR): ≤ 3 (19%) during the treatment period.
  5. Number of randomized patients per week: ≥ 3 patients.

SECONDARY OUTCOMES:
Visual Acuity | from baseline to end of follow-up at 7 months
  Change from baseline at 4 weeks, 1 month and 6 months:
  - Best Corrected Visual Acuity, distance and near vision (range 20/12.5 to <20/1000, higher score = better outcome)
Retinal Sensitivity | from baseline to end of follow-up at 7 months
  Change from baseline at 4 weeks,1 month and 6 months:
  - Mean retinal sensitivity (Macular Integrity Assessment, MAIA microperimetry - score: 0 dB to 36 dB, higher score = better outcome)
Fixation stability | from baseline to end of follow-up at 7 months
  Change from baseline at 4 weeks,1 month and 6 months:
  - Mean fixation stability (Macular Integrity Assessment, MAIA microperimetry - range 0.02 sq.deg. to 40.0 sq.deg., lowest score = better outcome)
Contrast Sensitivity | from baseline to end of follow-up at 7 months
  Change from baseline at 4 weeks, 1 month and 6 months:
  - Mean contrast sensitivity (Functional Acuity Contrast Test, FACT - range 0.48 cyc./deg. to 2.41 cyc./deg., higher score = better outcome)
Reading Speed | from baseline to end of follow-up at 7 months
  Change from baseline at 4 weeks,1 month and 6 months:
  - Mean reading speed (Minnesota Low Vision Reading test, MNREAD - range 0 word/minute to 280 word/minute, higher score = better outcome)
Quality of Life Scores | from baseline to end of follow-up at 7 months
  Change from baseline at 4 weeks,1 month and 6 months:
  - Quality of life scores (Veteran's Affairs Low Vision Questionnaire, VA-LVQ 48 - range -31.5 to +26.6, higher score = better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Krembil Research Institute/Toronto Western Hospital, Toronto, Ontario, Canada